CLINICAL TRIAL: NCT00683436
Title: A Multi-Center, Randomized, Blinded, Active and Placebo-Controlled, Crossover Study of the Efficacy and Safety of Two Doses of Adipiplon Bilayer Tablets in Primary Insomniacs
Brief Title: Efficacy and Safety Study of Adipiplon, Placebo and an Active Control in Primary Insomniacs
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Neurogen Corporation (Industry)
Responsible Party: Study Manager, Neurogen Corporation
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NG2-73-205
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2008-07-22 (Estimated); Status verified 2008-07

CONDITIONS: Primary Insomnia
Keywords: insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — adipiplon; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): adipiplon 6 mg
  Interventions: Drug: Adipiplon
- 2 (Experimental): adipiplon 9 mg
  Interventions: Drug: Adipiplon
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 4 (Experimental): Ambien CR 12.5 mg
  Interventions: Drug: Ambien CR

INTERVENTIONS:
Drug: Adipiplon — bilayer tablets 6 mg
  Arms: 1
Drug: Placebo — Placebo
  Arms: 3
Drug: Ambien CR — Ambien CR 12.5 mg
  Arms: 4
Drug: Adipiplon — bilayer tablets 9 mg
  Arms: 2

SUMMARY:
This will be a multi-center, randomized, blinded, comparative, placebo-controlled, 4 arm crossover study in patients with primary insomnia.

DETAILED DESCRIPTION:
Prospective patients will spend 2 nights in the sleep lab for baseline PSG assessments. Those who meet the protocol inclusion/exclusion criteria will return for four treatment periods with two consecutive nights in each. Study medication will be administered in the sleep laboratory 30 minutes before the patient's usual bedtime.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 21 and 64 years, inclusive;
* Have a body mass index (BMI) between 21 and 34 kg/m2, inclusive;
* Be a primary insomniac as defined by DSM-IV criteria; in particular difficulty with both sleep initiation and sleep maintenance;
* Have subjective Latency to Sleep Onset > 45 minutes;
* Have a mean habitual subjective TST of <6.5 hours;
* Have a TST of 240 - 420 minutes at each of two baseline PSGs;
* Have a mean LPS > 20min, with neither value <15 minutes and mean WASO > 40 minutes on baseline PSGs;
* Be in good general health as determined by a thorough medical history and physical examination (including vital signs), 12-lead ECG and clinical laboratory tests;
* Have clinical laboratory values within normal reference range or not clinically significantly abnormal as judged by the Principal Investigator;
* Be off any investigational drug for at least 30 days prior to screening;
* If the patient is a female of childbearing potential, she must be using an acceptable method of contraception, must have a negative serum pregnancy test at screening, and must have a negative urine pregnancy test before randomization.
* Female patients who have been surgically sterilized or have had a hysterectomy are eligible if they have a negative pregnancy test at screening;
* Be able to read, understand, and provide written/dated informed consent before enrolling in the study, and must be willing to comply with all study procedures.

Exclusion Criteria:

* Clinically significant unstable medical illness;
* Evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease;
* History of cancer other than basal cell carcinoma, squamous cell carcinoma of the skin or cancer in situ within 5 years of screening;
* Supine or sitting blood pressure > 140/90 mmHg at the screening or baseline visits;
* Heart rate >100 bpm at the screening or baseline visits;
* Within the past three years, clinically significant psychiatric illness, including chronic psychiatric illness or any Axis I condition;
* History or presence of chronic pain;
* History of epilepsy or serious head injury;
* Other than primary insomnia, a history of clinically significant sleep disorder including narcolepsy, parasomnia as an adult, circadian rhythm disorder, restless leg syndrome, or on the initial baseline PSG, sleep apnea [Apnea Hypopnea Index (AHI) >10] or Periodic Limb Movement Disorder [Periodic Limb Movement Arousal Index (PLMAI) > 10];
* Any condition that may affect drug absorption;
* Smokers who habitually smoke more than 10 cigarettes per day or smoke during the overnight hours;
* Travel across more than three time zones, an expected change in sleep schedules of 3 hours or more, or involvement in rotating shift work within 14 days prior to screening or during the study period;
* Self-report of napping ≥30 minutes more than 2 times per week within the last month;
* Any clinically significant abnormal finding on physical examination, vital signs, ECG, or clinical laboratory tests, as determined by the investigator. (The QTc interval must be ≤430 msec. for males and ≤450 msec for females);
* Known or suspected diagnosis of Acquired Immune Deficiency Syndrome, or previous or current positive result on human immunodeficiency virus antibody or antigen testing;
* History or laboratory finding of positive hepatitis B surface antigen or hepatitis C core antibody;
* History of allergies, or known sensitivity, hypersensitivity, or adverse reaction to any drug similar to adipiplon, including benzodiazepines, or zolpidem, zaleplon, zopiclone, or eszopiclone;
* Use of any psychotropic medications, including over-the-counter (OTC) and herbal products, that may affect sleep/wake function within one week or five half-lives (whichever is longer) prior to screening or need to use any of these medications at any time during the study;
* Pregnant or lactating females;
* Positive serum pregnancy test at screening or urine pregnancy test at baseline;
* Recent history (≤ one year) of alcohol or drug abuse, or current evidence of substance dependence or abuse as defined by DSM-IV criteria;
* Regular consumption of large amounts of xanthine-containing substances (i.e. more than 5 cups of coffee or equivalent amounts of xanthine-containing substances per day);
* Have eaten grapefruit or had grapefruit juice from baseline through the completion of study dosing;
* Self report of a usual consumption of more than 14 units of alcohol per week;
* Requiring the concomitant usage of any 3A4 inhibitors;
* Any prior exposure to adipiplon (formerly known as NG2-73).

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-10 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
The study will involve PSG measurement of sleep onset and maintenance. | two consecutive nights on each treatment

SECONDARY OUTCOMES:
The study will involve subjective measures of sleep and next day function. | two consecutive nights on each treatment

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Broward Research Group, Pembroke Pines, Florida
  - Miami Research Associates, South Miami, Florida
  - Neurotrials Research, Inc, Atlanta, Georgia
  - Sleep and Behavior Medicine Institute, Vernon Hills, Illinois
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - St. Luke's Hospital Sleep Medicine and Research Center, Chesterfield, Missouri
  - Clinilabs, Inc., New York, New York
  - Tri-State Sleep Disorders Center, Cincinnati, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma